CLINICAL TRIAL: NCT01522001
Title: Shared Care Rehabilitation After Acute Coronary Syndrome
Acronym: SHARED-REHAB
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Region MidtJylland Denmark (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: SHARED REHAB
Record Dates: First submitted 2012-01-26; First posted 2012-01-31 (Estimated); Last update posted 2015-05-29 (Estimated); Status verified 2012-09

CONDITIONS: Acute Coronary Syndrome; Myocardial Ischemia; Acute Myocardial Infarction: Rehabilitation Phase
Keywords: Acute Coronary Syndrome; Myocardial Ischemia; Shared Care; Rehabilitation; Community; Cardiac Rehabilitation; Hospital
MeSH Terms: conditions — Acute Coronary Syndrome; Myocardial Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hospital-based (No Intervention): * First visit at cardiac ambulatory approximately 14 days after discharge includes physician examination by cardiologist and counseling from nurse specialized in cardiac rehabilitation.
  * Dietary counseling with dietician
  * Exercise (1 hour, 2 timer pr week for 12 weeks)
  * Smoking cessation if smoker with educated smoking cessation instructor
  * Patient education and psychosocial support in 2 to 3 individual consultations with nurse specialized in cardiac rehabilitation
  * Examination by cardiologist 8-12 weeks after discharge.
- Shared care Model (Active Comparator): * First visit at cardiac ambulatory approximately 14 days after discharge includes examination by cardiologist and counseling from nurse specialized in cardiac rehabilitation.
  * Dietary counseling with dietician
  * Exercise (1 hour, 2 timer pr week for 12 weeks)
  * Smoking cessation if smoker with educated smoking cessation instructor
  * Patient education and psychosocial support in 2 individual consultations and 8 group based consultations with experienced nurse
  * Examination by the patient´s general practitioner 8-12 weeks after discharge.
  Interventions: Behavioral: Shared Care model

INTERVENTIONS:
Behavioral: Shared Care model — * First visit at cardiac ambulatory approximately 14 days after discharge includes physician examination by cardiologist and counseling from nurse specialized in cardiac rehabilitation.
  * Dietary counseling with dietician
  * Exercise (1 hour, 2 timer pr week for 12 weeks)
  * Smoking cessation if smoker with educated smoking cessation instructor
  * Patient education and psychosocial support in 2 individual consultations and 8 group based consultations with experienced nurse
  * Examination by the patient´s general practitioner 8-12 weeks after discharge.
  Arms: Shared care Model

SUMMARY:
Cardiac rehabilitation is an individual adapted multidisciplinary intervention for people suffering from Heart Disease. It involves;

* Dietary counseling,
* Exercise training,
* Psychosocial support,
* Physician
* smoking cessation
* Patient education

The purpose is quick and complete recovery and to reduce the chance of recurrence.

In Denmark people admitted with Acute Cardiac Disease is referred to a course of hospital based cardiac rehabilitation at discharge.

The Danish Municipal Reform of 2007 changed the responsibility of rehabilitation from the Regions, who runs the hospitals, to the municipalities.

Shared care is in this setting that elements of treatment are completed different places in Health Care.

The aim of this study is:

* to establish a shared care model for Cardiac rehabilitation following admission with Acute Coronary Syndrome and
* to compare this model to the existing hospital based cardiac rehabilitation after admission with Acute Coronary Syndrome.

Primary outcome is participation in cardiac rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Admission with Acute Coronary Syndrome
* Resident in district of Department of Cardiology, Aarhus University Hospital, Silkeborg or Viborg Hospital, part of the "Hospitalsenheden Midt" Viborg, Silkeborg, Skive, Hammel.
* Accept both models of cardiac rehabilitation
* written informed consent

Exclusion Criteria:

* Resident outside the district of Department of Cardiology, Aarhus University Hospital, Viborg Hospital or Silkeborg Hospital, part of "Hospitalsenheden Midt" (Viborg, Silkeborg, Skive, Hammel).
* Age 80 years or older
* Heart Failure (Ejection Fraction less than 40%)
* Severe Comorbidity
* Resuscitated and need of support from ergotherapist after discharge.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 212 (Actual)
Dates: Start 2011-10; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Participation in cardiac rehabilitation | 4 months
  Participation in cardiac rehabilitation is evaluated for each element. Participation is defined as at least 50% for each element.
  * Smoking cessation
  * Dietary counseling
  * Exercise training
  * Physician
  * Patient education
  * Psychosocial support
  Full participation is in 6 of 6 elements if smoker or 5/5 if non-smoker. Partial full participation is in 5/6 if smoker or 4/5 if non-smoker.

SECONDARY OUTCOMES:
Change of BMI and / or abdominal circumference | 4 and 12 months
24-hour Ambulatory Blood Pressure | 4 og 12 months
Blood Cholesterol values (Total, LDL, HDL) | 4 and 12 months
Fasting Blood glucose | 4 and 12 months
Exercise Capacity | 4 and 12 months
Lifestyle changes | 4 and 12 months
  Diet, Physical Activity, Smoking, Alcohol consumption.
Depression score | 4 and 12 months
  Estimated by Hospital Anxiety and Depression Scale
Compliance to pharmaceutical treatment | 4 and 12 months
Readmission | 4 and 12 months
  Total and cardiovascular
Change in Health Related Quality of Living | 4 and 12 months
  SF-12 HeartQoL EQ-5D
Difference in Health economic costs | 4 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Jannik B Bertelsen, MD, Principal Investigator — Hjertemedicinsk Afdeling B, Aarhus University Hospital
Locations (3):
- Denmark (3):
  - Silkeborg Hospital, Silkeborg, Region Midt
  - Aarhus University Hospital. Department of Cardiology and Medicine, Aarhus
  - Viborg Hospital, Hospital Unit of Viborg, Silkeborg, Hammel and Skive, Viborg

REFERENCES:
- [Derived] Bertelsen JB, Dehbarez NT, Refsgaard J, Kanstrup H, Johnsen SP, Qvist I, Christensen B, Sogaard R, Christensen KL. Shared care versus hospital-based cardiac rehabilitation: a cost-utility analysis based on a randomised controlled trial. Open Heart. 2018 Feb 7;5(1):e000584. doi: 10.1136/openhrt-2016-000584. eCollection 2018. PMID 29531754
- [Derived] Bertelsen JB, Refsgaard J, Kanstrup H, Johnsen SP, Qvist I, Christensen B, Christensen KL. Cardiac rehabilitation after acute coronary syndrome comparing adherence and risk factor modification in a community-based shared care model versus hospital-based care in a randomised controlled trial with 12 months of follow-up. Eur J Cardiovasc Nurs. 2017 Apr;16(4):334-343. doi: 10.1177/1474515116666781. Epub 2016 Sep 23. PMID 27566597